CLINICAL TRIAL: NCT04895202
Title: Swiss Study of the Impact of Mayzent (Siponimod) on Secondary Progressive Multiple Sclerosis Patients in a Long-term Non-interventional Study
Brief Title: Swiss Study of the Impact of Mayzent on SPMS Patients in a Long-term Non-interventional Study
Acronym: SWISSMASIA
Status: Terminated | Type: Observational
Why Stopped: Insufficient patient recruitment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312ACH01
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Secondary Progressive Multiple Sclerosis With Inflammatory Disease Activity
Keywords: SPMS; secondary progressive multiple sclerosis; Siponimod; active disease; inflammatory disease activity; disability progression
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — siponimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Siponimod: Patients administered Siponimod as per Swiss label
  Interventions: Other: Siponimod

INTERVENTIONS:
Other: Siponimod — Prospective observational cohort study. There is no treatment allocation. Patients administered siponimod as by swiss label, that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This study is a national, prospective, multicenter, non-interventional (observational) study with the aim to describe the impact of Siponimod treatment in a real-world SPMS population in Switzerland who are treated with Siponimod as per Swiss label.

DETAILED DESCRIPTION:
Primary data will be collected during an observational period of three years of Siponimod treatment. Additionally, medical history of participants will be collected including EDSS, MRI outcomes, relapses and previous medication to allow the estimation of Siponimod treatment effects on an individual basis. It is planned to include an optional blood draw for a later biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Adult patients with a documented diagnosis of SPMS with inflammatory disease activity who are going to be treated with Siponimod under routine medical care and in accordance with the Swiss label
3. Patient willing and able to complete the questionnaires

Exclusion Criteria:

1. Patients treated outside of the approved Swiss label for Siponimod
2. Prior treatment or already ongoing treatment with Siponimod
3. Use of investigational drugs during the study, OR within 3 months before enrollment, OR within 5 half-lives of investigational drug before enrollment, OR until the expected pharmacodynamic effect has returned to baseline, whichever is longer
4. Subjects who are not able to provide consent due to incapable judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SPMS population in Switzerland who are treated with Siponimod as per Swiss label
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change of expanded disability status scale (EDSS) | Baseline, month 36
  The EDSS score is a widely used tool for determining the degree of disability in MS at any point in time. The EDSS value is generated based on overall impression and individual scores of the following functional systems: cognition, mood, fatigue, vision, brain stem, upper extremities, lower extremities, bladder and bowel function, sexuality. This results in a scale from 0 (healthy) to 10 (death from MS)

SECONDARY OUTCOMES:
Proportion of patients with six month confirmed disability progression (CDP) by expanded disability status scale (EDSS) | month 36
  Disability progression based on the EDSS score is defined as a 1 point increase from baseline in patients with a baseline score of ≤ 5, or a 0.5 point increase in patients with a baseline score of ≥5.5. As part of a secondary endpoint to this study, the deterioration of the EDSS of ≥1 point (baseline EDSS ≤ 5) or 0.5 points (baseline EDSS ≥5.5) must be confirmed after 6 months. This is called 6-month confirmed progression (6M-CDPEDSS). EDSS values to confirm progression must not be determined during an attack. The maximum duration of an attack is limited to 90 days
Proportion of patients with six month confirmed disease progression by symbol digit modalities test (SDMT) | Up to 36 months
  The SDMT is a sensitive and specific test for examining attention, concentration and information processing speed, which are typically impaired in cognitively impaired MS patients.
  The patients receive an SDMT test sheet. At the beginning of this sheet there are 9 numbers paired with 9 associated individual symbols. Below that are further lines with symbols and empty boxes. The patients must now verbally assign the correct numbers to the symbols as quickly as possible. Exercise examples are given at the beginning of the test which are not taken into account when evaluating the test. The number of correctly assigned items within 90 seconds results into the test score. The total duration of the test is about 5 minutes.
  SDMT: ≥4.0-point confirmed worsening from baseline score sustained for at least 6 months respectively
Treatment effect of Siponimod on walking speed as measured by the timed 25 foot walk test (T25FWT) | Baseline, up to 36 months
  The T25-FW is an objective and quantitative test of the lower extremities (Motl et al., 2017). This stops the time in seconds that a patient needs to walk 25 feet (7.62 m). The patient should walk as quickly and safely as possible. This test is carried out twice in succession and the mean value of the time required is documented in seconds. An improvement or deterioration of 20% is seen as a clinical meaningful change (Motl et al., 2017).
Treatment effect of Siponimod on quality of life based on EQ-5D | Baseline, month 36
  The EQ-5D patient questionnaire is a generic multidimensional measuring instrument for describing health-related quality of life (EuroQol, 1999). The five domains mobility, ability to take care of oneself, everyday activities, pain / discomfort and anxiety / depression are considered. For the individual dimensions, the most appropriate answer from three given options is selected (1 = no problem, 2 = moderate problem, 3 = major problem). In addition, the patient marks the current state of health on a scale from 0 (worst-conceivable state of health) to 100 (best-conceivable state of health).
Treatment effect of Siponimod on fatigue measured by Fatigue Scale for Motor and Cognitive Functions (FSMC) | Baseline, month 36
  The FSMC is a patient questionnaire to clarify cognitive and motor fatigue, a typical symptom of MS (Penner et al., 2009). With the help of the FSMC, a cognitive, a motor, and a total score are determined. Increased scores indicate higher impairment caused by fatigue.
  A 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question.
Treatment effect of Siponimod on fatigue measured by Beck's depression inventory (BDI) | Baseline, month 36
  BDI is a patient questionnaire for measuring the severity of depression (Beck, 1972). Depression is a common symptom in MS and can cause fatigue. With the BDI test we assess the frequency of depression and its correlation to fatigue. This results in a scale from 0 to 63. The level of depression is evaluated according to the table below:
  * 0-13: no or minimal symptoms
  * 14-19: mild symptoms
  * 20-28: moderate symptoms
  * 29-63: severe depressive symptoms
Treatment effect of Siponimod on fatigue measured by Epworth sleepiness scale (ESS) questionnaire | Baseline, month 36
  ESS is a patient questionnaire to measure daytime sleepiness (Ibanez et al, 2017). Results of the ESS will allow to correlate whether observed fatigue might be attributed to daytime sleepiness. The level of sleepiness is evaluated according to the table below:
  0-5 Lower Normal Daytime Sleepiness 6-10 Higher Normal Daytime Sleepiness 11-12 Mild Excessive Daytime Sleepiness 13-15 Moderate Excessive Daytime Sleepiness 16-24 Severe Excessive Daytime Sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceiticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Switzerland (6):
  - Novartis Investigative Site, Zug, Canton of Zug
  - Novartis Investigative Site, Zurich, Canton of Zurich
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Winterthur

IPD SHARING:
Plan to Share IPD: No